CLINICAL TRIAL: NCT01357616
Title: Comparison of Efficacy and Safety of Brinzolamide/Timolol Fixed Combination (AZARGA™) vs Brinzolamide (AZOPT®) and Timolol in Chinese Subjects With Open-Angle Glaucoma or Ocular Hypertension
Brief Title: Fixed Combination Brinzolamide 1%/Timolol 0.5% Versus Brinzolamide 1% + Timolol 0.5% in Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C-08-076
Record Dates: First submitted 2011-05-18; First posted 2011-05-20 (Estimated); Results first posted 2014-03-13 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-03

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
Keywords: Glaucoma; Open-angle glaucoma; Ocular hypertension; OAG; OH
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma | interventions — brinzolamide; Timolol; Azarga; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZARGA (Experimental): Brinzolamide 1% / Timolol 0.5% fixed combination ophthalmic suspension, 1 drop in the affected eye(s) dosed twice daily (9AM and 9PM) for 8 weeks. Both eyes were dosed unless there was a potential safety issue to the patient in the opinion of the Investigator.
  Interventions: Drug: Brinzolamide 1% / Timolol 0.5% fixed combination ophthalmic suspension
- AZOPT + Timolol (Active Comparator): Brinzolamide 1% ophthalmic suspension, 1 drop instilled in the affected eye(s), followed by Timolol 0.5% ophthalmic solution, 1 drop instilled in the affected eye(s). Approximately 10 minutes separated the 2 instillations. The study drugs were instilled twice daily (9AM and 9PM) for 8 weeks. Both eyes were dosed unless there was a potential safety issue to the patient in the opinion of the Investigator.
  Interventions: Drug: Brinzolamide 1% ophthalmic suspension; Drug: Timolol 0.5% ophthalmic solution

INTERVENTIONS:
Drug: Brinzolamide 1% / Timolol 0.5% fixed combination ophthalmic suspension
  Other Names: AZARGA™
  Arms: AZARGA
Drug: Brinzolamide 1% ophthalmic suspension
  Other Names: AZOPT®
  Arms: AZOPT + Timolol
Drug: Timolol 0.5% ophthalmic solution
  Other Names: TIMOLOL
  Arms: AZOPT + Timolol

SUMMARY:
The purpose of this study was to compare the intraocular pressure (IOP)-lowering efficacy and safety of AZARGA™ (Brinzolamide 1%/Timolol 0.5% Ophthalmic Suspension), dosed twice daily versus AZOPT® (Brinzolamide 1% Ophthalmic Suspension) and Timolol 0.5% Ophthalmic Solution, each dosed twice daily, in Chinese patients with open-angle glaucoma or ocular hypertension who were insufficiently responsive to monotherapy.

DETAILED DESCRIPTION:
The study consisted of 2 sequential phases. Phase I was the Screening/Eligibility Phase, with a Screening Visit followed by an Eligibility Visit. Phase II was the treatment phase and included Week 1, Week 2, Week 4, and Week 8 visits. Eligible subjects were randomized in a 1:1 ratio to receive Brinzolamide 1%/Timolol 0.5% or Brinzolamide 1% plus Timolol 0.5% two times a day for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with open angle glaucoma and/or ocular hypertension and not sufficiently responsive to monotherapy.
* Meet qualifying IOP criteria in at least 1 eye, including 21-35 mmHg at the Eligibility visit.
* Willing to sign an Informed Consent form.
* Contact lens wearer who is willing to remove lenses before instillation of study medication and wait a minimum of 15 minutes following drug instillation before re-inserting the lenses.
* Able to discontinue use of current IOP-lowering medications per the minimum washout period.
* Other protocol-specific inclusion criteria may apply.

Exclusion Criteria:

* Women of childbearing potential if pregnant, test positive for pregnancy at Screening/Enrollment visit, breastfeeding, or not in agreement to use adequate birth control methods to prevent pregnancy throughout the study.
* Diagnosed with any form of glaucoma other than open-angle glaucoma and/or ocular hypertension.
* Diagnosed with severe central visual field loss in either eye.
* History of chronic, recurrent, or severe ocular infection, inflammatory eye disease in either eye.
* History of ocular trauma within the past 6 months in either eye.
* Current ocular infection or ocular inflammation within the past 3 months in either eye.
* Ocular laser surgery within the past 3 months.
* Intraocular surgery within the past 3 months.
* Best-corrected visual acuity score worse than 55 ETDRS letters read (equivalent to approximately 20/80 Snellen, 0.60 logMAR or 0.25 decimal).
* History of, or current clinically relevant or progressive retinal disease in either eye.
* History of, or current other severe ocular pathology (including severe dry eye) in either eye, that would preclude the administration of a topical carbonic anhydrase inhibitor (CAI) or beta-blocker.
* Any abnormality preventing reliable applanation tonometry.
* History of, or current condition or disease that would preclude the safe administration of a topical beta blocker or topical beta-adrenergic blocking agent.
* History of spontaneous or current hypoglycemia or uncontrolled diabetes.
* History of severe or serious hypersensitivity to CAIs, beta-blockers, or to any components of the study medication.
* Less than 30 days stable dosing regimen before the Screening Visit of any medications or substances administered by any route and used on a chronic basis that may have affected IOP.
* Recent use of high-dose salicylate therapy.
* Anticipated use of any additional topical or systemic ocular hypotensive medication during the study.
* Not safely able to discontinue all glucocorticoid medications administered by any route.
* Currently on therapy or have been on therapy with another investigational agent within 30 days prior to the Screening Visit.
* History of, or current evidence of severe illness or any other conditions which would, in the opinion of the Investigator, make the subject unsuitable for the study.
* Other protocol-specific exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2010-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mandy Ye, MS, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 13 study centers located in China.
Pre-assignment Details: This reporting group includes all enrolled subjects.
Groups:
- AZOPT + TIMOLOL: Brinzolamide 1% ophthalmic suspension and Timolol 0.5% ophthalmic solution, 1 drop of each component instilled in the affected eye(s), waiting approximately 10 minutes between instillation of the 2 drops. Study drugs were instilled twice daily (9AM and 9PM) for 8 weeks.
Period: Overall Study
Arm/Group | AZARGA | AZOPT + TIMOLOL
Started | 166 | 162
Completed | 156 | 153
Not Completed | 10 | 9
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 4 | 3
Not completed — Protocol Violation | 0 | 2
Not completed — Inadequate Control of IOP | 1 | 2
Not completed — Decision Unrelated to Adverse Event | 3 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: This reporting group includes all subjects who received study medication, satisfied pre-randomization inclusion/exclusion criteria and completed at least 1 scheduled on-therapy study visit.
Groups:
- Total: Total of all reporting groups
Arm/Group | AZARGA | AZOPT + TIMOLOL | Total
Number analyzed (Participants) | 157 | 155 | 312
Age, Customized [Number; unit: participants]
  <65 Years | 148 | 135 | 283
  ≥65 Years | 9 | 20 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 72 | 141
  Male | 88 | 83 | 171

OUTCOME MEASURES:

1. Primary Outcome: Mean Diurnal IOP Change From Baseline at Week 8
Description: Mean diurnal IOP change from baseline at Week 8 (ie, the subject IOP change from baseline averaged over the 9 AM, 11AM and 5 PM time points at Week 8) was measured by Goldmann applanation tonometry. One eye from each subject was chosen as the study eye, and only data for the study eye were used for the efficacy analysis. A higher IOP (fluid pressure inside the eye) can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage). A more negative change indicates a greater improvement..
Time Frame: Baseline, Week 8
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Deviation); unit: millimeters mercury (mmHg)
Arm/Group | AZARGA | AZOPT + Timolol
Number analyzed (Participants) | 157 | 155
millimeters mercury (mmHg) | -6.84 (3.557) | -6.00 (2.934)

2. Secondary Outcome: Mean IOP Change From Baseline at 9 AM
Description: Mean IOP change from baseline at 9 AM was measured by Goldmann applanation tonometry. One eye from each subject was chosen as the study eye, and only data for the study eye were used for the efficacy analysis. A higher IOP (fluid pressure inside the eye) can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage). A more negative change indicates a greater improvement.
Time Frame: Baseline, Up to Week 8
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Deviation); unit: mmHg
Arm/Group | AZARGA | AZOPT + Timolol
Number analyzed (Participants) | 157 | 155
mmHg
  Change from baseline at Week 2 | -6.9 (3.62) | -6.5 (3.43)
  Change from baseline at Week 4 | -7.3 (3.42) | -6.4 (3.11)
  Change from baseline at Week 8 | -6.7 (3.97) | -6.2 (3.30)

3. Secondary Outcome: Mean IOP Change From Baseline at 11 AM
Description: Mean IOP change from baseline at 11 AM was measured by Goldmann applanation tonometry. One eye from each subject was chosen as the study eye, and only data for the study eye were used for the efficacy analysis. A higher IOP (fluid pressure inside the eye) can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage). A more negative change indicates a greater improvement.
Time Frame: Baseline, Up to Week 8
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Deviation); unit: mmHg
Arm/Group | AZARGA | AZOPT + Timolol
Number analyzed (Participants) | 157 | 155
mmHg
  Change from baseline at Week 2 | -7.5 (3.19) | -6.8 (3.07)
  Change from baseline at Week 4 | -7.6 (3.46) | -6.8 (3.06)
  Change from baseline at Week 8 | -7.4 (3.92) | -6.5 (3.57)

4. Secondary Outcome: Mean IOP Change From Baseline (5 PM) at Week 8
Description: Mean IOP change from baseline (5 PM) at Week 8 was measured by Goldmann applanation tonometry. One eye from each subject was chosen as the study eye, and only data for the study eye were used for the efficacy analysis. A higher IOP (fluid pressure inside the eye) can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage). A more negative change indicates a greater improvement.
Time Frame: Baseline, Week 8
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Deviation); unit: mmHg
Arm/Group | AZARGA | AZOPT + Timolol
Number analyzed (Participants) | 157 | 155
mmHg | -6.3 (3.99) | -5.1 (3.34)

ADVERSE EVENTS:
Time Frame: Adverse Events (AE) were collected for the duration of the study (2 years, 2 months). An AE was defined as any untoward medical occurrence in a subject who was administered a study treatment, regardless of causal relationship with the treatment.
Description: Of the 328 enrolled, 1 subject did not receive study medication. This reporting group includes all subjects who were randomized and received study medication (327). Reports of AEs were obtained through solicited and spontaneous comments from the study subjects, and through observations by the study Investigator as outlined in the study protocol.
Groups:
- AZARGA (Test Group): Brinzolamide 1% / Timolol 0.5% fixed combination ophthalmic suspension, 1 drop in the affected eye(s) dosed twice daily (9AM and 9PM) for 8 weeks.
  Brinzolamide 1% / Timolol 0.5% fixed combination ophthalmic suspension
- AZOPT + TIMOLOL (Control Group): Brinzolamide 1% ophthalmic suspension and Timolol 0.5% ophthalmic solution, 1 drop of each component instilled in the affected eye(s), waiting approximately 10 minutes between instillation of the 2 drops. Study drugs were instilled twice daily (9AM and 9PM) for 8 weeks.
  Brinzolamide 1% ophthalmic suspension and Timolol 0.5% ophthalmic solution
Arm/Group | AZARGA (Test Group) | AZOPT + TIMOLOL (Control Group)
Serious Adverse Events (participants affected / at risk) | 1/165 | 0/162
Other Adverse Events (participants affected / at risk) | 14/165 | 10/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZARGA (Test Group) (N=165) | AZOPT + TIMOLOL (Control Group) (N=162)
Benign neoplasm of thymus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZARGA (Test Group) (N=165) | AZOPT + TIMOLOL (Control Group) (N=162)
Heart rate decreased (Investigations) | 14 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.